CLINICAL TRIAL: NCT01983826
Title: Dietary Nitrates and Vascular Function in Patients With Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Darren P Casey, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 201307745; 13GRNT16490002 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2013-10-28; First posted 2013-11-14 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Peripheral Artery Disease
Keywords: nitrates; blood flow; vascular function; exercise
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity | interventions — sodium nitrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Nitrate (Experimental): Sodium Nitrate (1g/day) for 8 weeks
  Interventions: Dietary Supplement: Sodium Nitrate
- Placebo capsule (Placebo Comparator): Microcrystalline cellulose (daily) for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Sodium Nitrate — Sodium Nitrate (1g/day) for 8 weeks
  Arms: Sodium Nitrate
Other: Placebo — Microcrystalline cellulose (daily) for 8 weeks
  Arms: Placebo capsule

SUMMARY:
The overarching question addressed in the current project is: Does dietary nitrate supplementation (8 weeks) improve physiological function in patients with peripheral arterial disease (PAD)? The investigators will specifically address whether dietary nitrate supplementation enhances blood vessel function, blood pressure regulation, and exercise capacity. The proposed project uses an array of clearly defined measurements which will allow investigators to quantify blood vessel function (vasodilator responsiveness and arterial stiffness), blood pressure (variability and responsiveness to stress), and functional capacity before and after 8 weeks of dietary supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Documented peripheral artery disease
* Ankle-Brachial Index (ABI) < or = to 0.90

Exclusion Criteria:

* Non-atherosclerotic vascular disease
* Critical limb ischemia
* Active ischemic ulceration
* Recent (within one year) revascularization
* Symptomatic coronary artery disease (angina pectoris)
* Heart failure
* Resting systolic blood pressure > 180 mmHg or diastolic pressure > 100 mmHg
* Hypotension (resting systolic BP < 90 mmHg)
* Smoking or history of smoking within past one year
* Use of phosphodiesterase V inhibitor drugs
* Women with history of hormone replacement therapy within the past 6 months

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren P Casey, Ph.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Hughes WE, Treichler DP, Ueda K, Bock JM, Casey DP. Sodium nitrate supplementation improves blood pressure reactivity in patients with peripheral artery disease. Nutr Metab Cardiovasc Dis. 2022 Mar;32(3):710-714. doi: 10.1016/j.numecd.2021.12.002. Epub 2021 Dec 8. PMID 35090799

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Nitrate (NaNO3): Subjects randomized to this group took Sodium Nitrate capsules (1g/day) for 8 weeks
- Placebo: Subjects randomized to this group took a daily Placebo capsule (Microcrystalline cellulose) for 8 weeks
Period: Overall Study
Arm/Group | Sodium Nitrate (NaNO3) | Placebo
Started | 13 | 8
Completed | 13 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Nitrate (NaNO3) | Placebo | Total
Number analyzed (Participants) | 13 | 8 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 11 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (9) | 69 (10) | 72 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 7 | 2 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 8 | 21
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (5.9) | 28.1 (3.6) | 28.8 (5.1)
Ankle-brachial index (ABI) [Mean (Standard Deviation); unit: ratio] — Ankle Brachial Index (ABI) is the ratio of the blood pressure in the lower legs to the blood pressure in the arms. Compared to the arm, lower blood pressure in the leg may be a symptom of peripheral artery disease (PAD) or a blockage in the leg. Ranges for ABI values are:
  No blockage (1.0 to 1.4)
  Borderline blockage (0.91 to 0.99). An ankle-brachial index number is this range indicates that you have borderline PAD.
  PAD (less than 0.90). An ankle-brachial index number in this range is considered abnormal and indicates a diagnosis of PAD.
  ratio | 0.76 (0.21) | 0.81 (0.14) | 0.78 (0.18)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 136 (15) | 132 (13) | 135 (14)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 72 (9) | 77 (10) | 74 (10)

OUTCOME MEASURES:

1. Primary Outcome: Change in Vasodilator Capacity
Description: Forearm and calf blood flow will be measured independently by venous occlusion plethysmography using mercury-in-silastic strain gauges. Plethysmographic measurements will be made at rest and following 5 minutes of ischemia (reactive hyperemia) of the distal limb (forearm and calf). Peak blood flow will be determined as the highest flow recorded during the post deflation period. Total blood flow will be measured as the area under the time-curve after resting flow is subtracted. Vascular conductance will be calculated using blood flow/mean arterial pressure (via finger plethysmograph).
Time Frame: Pre and post 8 weeks of dietary nitrate supplementation
Population: Calf blood flow measures were only performed in 11 of the subjects in the NaNO3 group and 7 of the subjects in the Placebo group.
Measure: Mean (Standard Deviation); unit: ml/100ml tissue/min
Groups:
- Sodium Nitrate (NaNO3) Pre: Subjects randomized to this group took Sodium Nitrate capsules (1g/day) for 8 weeks Values reflect pre intervention measures
- Sodium Nitrate (NaNO3) Post: Subjects randomized to this group took Sodium Nitrate capsules (1g/day) for 8 weeks Values reflect post intervention measures
- Placebo - Pre: Subjects randomized to this group took a daily Placebo capsule (Microcrystalline cellulose) for 8 weeks Values reflect pre intervention measures
- Placebo - Post: Subjects randomized to this group took a daily Placebo capsule (Microcrystalline cellulose) for 8 weeks Values reflect post intervention measures
Arm/Group | Sodium Nitrate (NaNO3) Pre | Sodium Nitrate (NaNO3) Post | Placebo - Pre | Placebo - Post
Number analyzed (Participants) | 13 | 13 | 8 | 8
ml/100ml tissue/min
  Peak forearm Blood Flow | 16.2 (6.6) | 16.4 (4.2) | 16.5 (5.2) | 14.2 (7.2)
  Peak calf Blood Flow: number analyzed (Participants) | 11 | 11 | 7 | 7
  Peak calf Blood Flow | 11.6 (4.9) | 14.1 (5.1) | 13.1 (3.5) | 11.9 (3.7)

2. Primary Outcome: Change in Arterial Stiffness
Description: ECG gated arterial waveforms will be obtained via applanation tonometry from the carotid and femoral arteries. The pulse wave velocity (PWV; index of arterial stiffness) will be determined between the carotid and femoral measurement sites (cfPWV). The time (t) between the feet of recorded pressure waves will be determined as the mean of 10 consecutive cardiac cycles. PWV is calculated from the distance (D; meters) between measurement points and the measured time delay (t): PWV = D/Δt (m/s).
Time Frame: Pre and post 8 weeks of dietary nitrate supplementation
Population: We were only able to obtain quality PWV measures in 11 subjects in the sodium nitrate group and 6 in the placebo group.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Sodium Nitrate (NaNO3) Pre | Sodium Nitrate (NaNO3) Post | Placebo - Pre | Placebo - Post
Number analyzed (Participants) | 11 | 11 | 6 | 6
m/sec | 13.8 (3.4) | 12.8 (2.9) | 10.5 (3.1) | 11.0 (3.7)

3. Primary Outcome: Change in Functional Capacity - Distance Walked in 6 Minutes
Description: 6-minute walk tests will be performed before and after treatment to assess functional capacity. The main comparisons will be changes distance walked in 6 minutes after 8 weeks of dietary nitrate supplementation.
Time Frame: Pre and post 8 weeks of dietary nitrate supplementation
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Sodium Nitrate (NaNO3) Pre | Sodium Nitrate (NaNO3) Post | Placebo - Pre | Placebo - Post
Number analyzed (Participants) | 13 | 13 | 8 | 8
meters | 387 (90) | 425 (82) | 423 (56) | 427 (66)

ADVERSE EVENTS:
Arm/Group | Sodium Nitrate (NaNO3) Pre | Sodium Nitrate (NaNO3) Post | Placebo - Pre | Placebo - Post
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No